CLINICAL TRIAL: NCT06701708
Title: Exploratory Study on Artifact Denoising of Cerebral Blood Flow and EEG Data in Ambulance Settings
Status: Not yet recruiting | Type: Observational
Sponsor: Pusan National University Yangsan Hospital (Other)
Responsible Party: Principal Investigator, Yong-il Shin, Professor, Pusan National University Yangsan Hospital
Other Study IDs: 11-2024-058
Record Dates: First submitted 2024-11-20; First posted 2024-11-22 (Actual); Last update posted 2024-11-22 (Actual); Status verified 2024-11

CONDITIONS: Normal; EEG; FNIRS

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Normal
  Interventions: Other: Participants are not assigned to interventions based on a protocol.

INTERVENTIONS:
Other: Participants are not assigned to interventions based on a protocol. — Participants are not assigned to interventions based on a protocol.

SUMMARY:
The purpose is to assess the extent of digital noise occurring during the measurement of cerebral blood flow and EEG in healthy adults within an ambulance setting and to explore the possibility of identifying and correcting abnormal patterns.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults aged 19 to 80 years.
* Individuals without chronic diseases (e.g., Stage 2 hypertension, cardiovascular disease, chronic kidney disease, chronic pulmonary disease, etc.).
* Individuals without mental health disorders (e.g., depression, schizophrenia, etc.).
* Individuals not taking medications that could affect cerebral hemodynamics, such as antihypertensives, anticoagulants, antiplatelets, antidepressants, etc.

Individuals who can read and understand the participant information and consent form and have sufficient language ability to respond to questionnaires.

- Individuals who voluntarily decide to participate in the clinical study, provide written consent on the participant consent form, and are able to participate throughout the entire duration of the clinical study.

Exclusion Criteria:

* Individuals who have experienced head trauma in the past 6 months.
* Individuals with ongoing severe chronic diseases (e.g., heart failure, chronic kidney disease, chronic pulmonary disease, etc.).
* Individuals with severe mental health disorders such as schizophrenia, severe depression, bipolar disorder, etc.
* Individuals currently taking medications that may affect the study (e.g., antihypertensives, anticoagulants, antiplatelets, antidepressants, etc.).
* Individuals who have participated in a clinical trial and taken experimental drugs within the past 30 days.
* Women who are pregnant or breastfeeding.
* Individuals who have undergone major surgery in the past 6 months.
* Individuals with acute infections or inflammatory diseases.
* Individuals with cognitive impairment or dementia.
* Individuals with neurological disorders.
* Individuals who lack understanding of the study procedures or who have not voluntarily consented to participate.
* Individuals with clinically significant findings that the study principal investigator or responsible medical personnel determines to be inappropriate for participation in this study.

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Normal individual
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2024-12-01 (Estimated); Primary Completion 2024-12-01 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Electroencephalography (EEG) signals in the ambulance | 10 minutes by boarding an ambulance in driving
  Electroencephalography (EEG) is used for measurement. Electroencephalography (EEG) is a non-invasive technique used to record the electrical activity of the brain through electrodes placed on the scalp. These electrodes detect and amplify signals generated by the synchronous activity of neurons, particularly in the cerebral cortex. EEG provides a real-time measure of brain activity with high temporal resolution, typically capturing signals in the range of 1-100 Hz.

SECONDARY OUTCOMES:
Functional Near-Infrared Spectroscopy(fNIRS) signals in the ambulance | 10 minutes by boarding an ambulance in driving
  Functional Near-Infrared Spectroscopy (fNIRS) is a non-invasive optical imaging technique used to measure changes in brain activity by detecting hemodynamic responses associated with neural activity. It relies on the absorption properties of near-infrared light, which penetrates the scalp and skull to assess oxygenated (HbO) and deoxygenated (HbR) hemoglobin levels in cortical regions.

IPD SHARING:
Plan to Share IPD: No